CLINICAL TRIAL: NCT06482437
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of NMD670 Over 21 Days in Ambulatory Adult Patients With Type 1 and Type 2 Charcot-Marie-Tooth Disease
Brief Title: Safety and Efficacy of NMD670 in Adult Patients With Type 1 and Type 2 Charcot-Marie-Tooth Disease
Acronym: SYNAPSE-CMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NMD Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMD670-02-0003
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NMD670 (Experimental)
  Interventions: Drug: NMD670
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NMD670 — Tablets taken twice daily for 21 days
  Arms: NMD670
Drug: Placebo — Tablets taken twice daily for 21 days
  Arms: Placebo

SUMMARY:
This Phase 2a study aims to evaluate the efficacy, safety and tolerability of NMD670 vs placebo administered twice a day (BID) for 21 days in ambulatory adult patients with Charcot-Marie-Tooth disease type 1 and type 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be 18 to 70 years inclusive at the time of signing the ICF.
* Diagnosis of CMT type 1 or 2 confirmed by genetic testing.
* Body mass index between 18 and 35 kg/m2, inclusive, at screening, and with a minimum weight of 40 kg
* Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Participant is capable of and has given signed informed consent

Exclusion Criteria:

* Participants with other significant disease that may interfere with the interpretation of study data (e.g., other neuromuscular diseases) and/or ability to complete the tests, in the opinion of the Investigator.
* Participants with laboratory test result abnormalities at screening considered clinically significant by the Investigator.
* Participants who have received treatment with another IMP within 30 days (or 5 half-lives of the medication, whichever is longer) prior to day 1.
* Participants with history of poor compliance with relevant therapy in the opinion of the Investigator.
* Female participants who plan to become pregnant during the study or are currently pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline to day 21 in 6-minute walk test total distance for NMD670 vs placebo | Baseline to day 21

SECONDARY OUTCOMES:
Change from baseline to day 21 in CMT Functional Outcome Measure Total Score and Individual Items for NMD670 vs placebo | Baseline to day 21
  CMT Functional Outcome Meausre is a 12-item scale. Scale goes from 0-100 and a higher score indicates worse symptomatology
Change from baseline to day 21 in the time to complete the 10MW/RT for NMD670 vs placebo | Baseline to day 21
Change from baseline to day 21 in 6-minute walk test fatigue index for NMD670 vs placebo | Baseline to day 21
Change from baseline to day 21 in Overall Neuropathy Limitation Scale total score and individual items for NMD670 vs placebo | Baseline to day 21
  The Overall Neuropathy Limitation Scale consists of an arm and a leg scale. Scale goes from 0-12 and a higher score indicates worse symptomatology
Change from baseline to day 21 in CMT Health Index total score and individual domains for NMD670 vs placebo | Baseline to day 21
  The CMT Health Index has 18 domains. Scale goes from 0-100 and a higher score indicates worse symptomatology
Change from baseline to day 21 in SF-36 total score and individual domains for NMD670 vs placebo | Baseline to day 21
  The SF-36 has 8 domains. Scale goes from 0-100 and a lower score indicates worse symptomatology
Change from baseline to day 21 in jitter and blocking for NMD670 vs placebo | Baseline to day 21
Incidence of treatment emergent adverse events | Over 21 days of dosing
  Summarised per treatment
Incidence of serious treatment emergent adverse events | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on physical examinations | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on safety laboratory parameters | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant vital signs abnormalities | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant ECG abnormalities | Over 21 days of dosing
  Summarised per treatment
Incidence of Suicidal Ideation or Suicidal Behavior | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on opthalmological examinations | From screening (day -28 to day -1) until follow up (day 28)]
  Summarised per treatment
Proportion of participants with clinically meaningful change from baseline in CMT-FOM total score and individual items for NMD670 vs placebo | Baseline to day 21
Proportion of participants with clinically meaningful change from baseline in 10MW/RT for NMD670 vs placebo | Baseline to day 21
Proportion of participants with clinically meaningful change from baseline in ONLS total score for NMD670 vs placebo | Baseline to day 21
Proportion of participants with clinically meaningful change from baseline in CMT-HI total score and individual domains for NMD670 vs placebo | Baseline to day 21
Proportion of participants with clinically meaningful change from baseline in SF-36 total score and individual domains for NMD670 vs placebo | Baseline to day 21

CONTACTS AND LOCATIONS:
Locations (19):
- United States (8):
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - Mass General Neurology, Boston, Massachusetts
  - NextGen Precision Health, Columbia, Missouri
  - Columbia University Medical Center, New York, New York
  - University of Rochester Neuromuscular Disease Center, Rochester, New York
  - OSU Department of Neurology Division of Neuromuscular Diseases, Columbus, Ohio
  - National Neuromuscular research Institute, PLLC, Austin, Texas
  - Providence Medical Research Center, Spokane, Washington
- Belgium (2):
  - University Hospitals Leuven, Department of Neurology, Leuven
  - CHR de la Citadelle- Site Citadelle Neurolgie Boulevard du 12eme de Ligne 1, Liège
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Department of Neurology, Copenhagen
- France (5):
  - CHU Marseille, Reference centre for neuromuscular diseases and ALS Department of Neuromuscular Diseases, Marseille
  - Laboratoire d'Explorations Fonctionnelles, CHU Nantes, Nantes
  - Centre Hospitalier Universitaire De Nice, Nice
  - Institut de Myologie Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Bicêtre University Hospital, Paris
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No